CLINICAL TRIAL: NCT04813016
Title: Comparative Study Between Intraperitoneal Administration of Either Bupivacaine and Tramadol Versus Bupivacaine and Dexmedetomedine for Analgesia After Abdominal Laparoscopic Cancer Surgeries. A Prospective Randomized Pilot Study
Brief Title: Intraperitoneal Tramadol Versus Dexmedetomedine for Analgesia After Abdominal Laparoscopic Cancer Surgeries
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: National Cancer Institute, Egypt (Other)
Responsible Party: Principal Investigator, Ehab Hanafy Shaker, Assistant professor of Anesthesia, intensive care and pain releif, National Cancer Institute, Egypt
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: intraperitoneal analgesia
Record Dates: First submitted 2021-03-20; First posted 2021-03-24 (Actual); Last update posted 2022-06-02 (Actual); Status verified 2022-06

CONDITIONS: Analgesia
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Early tramal/bupivacaine (Active Comparator): patients received 50 ml of isotonic aqueous solution (PH 7.45) of tramadol 150mg mixed with bupivacaine 0.25% immediately before creation of a pneumoperitoneum and placement of the first two trocars before starting the surgery.
  Interventions: Drug: Tramal 2; Drug: Dexmedetomidine 1; Drug: dexmedetomidine 2
- Late tramal/bupivacaine (Active Comparator): patients received 50ml of isotonic aqueous solution (PH 7.45) of tramadol 150mg mixed with bupivacaine 0.25% after completion of surgery and before trocars removal.
  Interventions: Drug: Tramal 1; Drug: Dexmedetomidine 1; Drug: dexmedetomidine 2
- Early dexmedetomedine/bupivacaine (Active Comparator): patients received 50ml of isotonic aqueous solution (PH 7.45) of dexmedetomedine(1µ/kg) mixed with bupivacaine 0.25% before creation of a pneumoperitoneum and placement of the first two trocars before the start of surgery.
  Interventions: Drug: Tramal 1; Drug: Tramal 2; Drug: dexmedetomidine 2
- Late dexmedetomedine/bupivacaine (Active Comparator): patients received 50ml of isotonic aqueous solution (PH 7.45) of dexmedetomedine(1µ/kg) mixed with bupivacaine 0.25% after completion of surgery and before trocars removal.
  Interventions: Drug: Tramal 1; Drug: Tramal 2; Drug: Dexmedetomidine 1

INTERVENTIONS:
Drug: Tramal 1 — Early intraperitoneal injection of tramal and bupivacaine
  Other Names: Early tramal
  Arms: Early dexmedetomedine/bupivacaine; Late dexmedetomedine/bupivacaine; Late tramal/bupivacaine
Drug: Tramal 2 — Late intraperitoneal injection of tramal and bupivacaine
  Other Names: Late tramal
  Arms: Early dexmedetomedine/bupivacaine; Early tramal/bupivacaine; Late dexmedetomedine/bupivacaine
Drug: Dexmedetomidine 1 — Early intraperitoneal injection of dexmedetomidine and bupivacaine
  Other Names: Early Dexmedetomidine
  Arms: Early tramal/bupivacaine; Late dexmedetomedine/bupivacaine; Late tramal/bupivacaine
Drug: dexmedetomidine 2 — Late intraperitoneal injection of dexmedetomedine and bupivacaine
  Other Names: Late Dexmedetomidine
  Arms: Early dexmedetomedine/bupivacaine; Early tramal/bupivacaine; Late tramal/bupivacaine

SUMMARY:
Multiple modalities for postoperative analgesia after laparoscopic procedures has been used, of them intraperitoneal route (IP) was used to decrease the analgesic requirements. Both early and late bupivacaine and tramadol versus bupivacaine and dexmedetomedine will be tried to choose which is having a better analgesic profile.

DETAILED DESCRIPTION:
Recently laparoscopic procedures have become popular and familiar to both surgeons and anesthetists. They have many advantages such as rapid postoperative recovery, low postoperative complication rates, early mobilization, and early home discharge; consequently reduce hospital stay and costs. Although previous studies have been shown that laparoscopy is associated with less pain than laparotomy, it is not totally pain free. Some laparoscopic procedures for abdominal cancer surgeries has shown that there may be more intense pain and greater analgesic requirements in the immediate postoperative period than after open laparotomy.

Thoroughly understanding the difference of pain generators in laparotomy than in laparoscopy gave some ideas helping in the control of each of them. While laparotomy results mainly in parietal pain, visceral pain remains predominantly in patients after laparoscopic surgeries resulting from the stretching of intra-abdominal cavity, peritoneal inflammation and phrenic nerve irritation caused by residual carbon dioxide in the peritoneal cavity resulting in postoperative abdominal and shoulder pain after laparoscopy. Hence, Intraperitoneal (IP) administration of some drugs can be effective for pain relief after laparoscopic surgery. The results have been variable as the published studies are heterogeneous and often lack appropriate controls. For that, no definitive conclusion can yet be made regarding its value and effectiveness.

The α2-adrenergic agonist provides excellent sedation, anxiolysis, analgesia and sympatholysis. Of them, dexmedetomidine has become one of the frequently used drugs in anaesthesia aiming to its hemodynamic, sedative, anxiolytic, analgesic, neuroprotective and anaesthetic sparing effect. In addition, the high selectivity of dexmedetomidine to α2- receptors favored its widespread use in regional anaesthesia practice and local nerve blocks techniques.

As noradrenergic neurons descending through the dorso-lateral funiculus from the brainstem to the dorsal horn significantly contribute in the modulation of pain by controlling impulse transmission (descending inhibitory pathway). Adrenergic agonists, such as dexmedetomedine, possess significant antinociceptive activity by a central action on the brainstem and a spinal action on the substantia gelatinosa of the dorsal horn.

Tramadol is a synthetic opioid pain medication used to treat moderate to moderately severe pain. It exerts its analgesic effects through a variety of different targets on the noradrenergic, serotoninergic and opioid receptors systems. It also exists as a racemic mixture, the positive enantiomer inhibits serotonin reuptake while the negative enantiomer inhibits noradrenaline re-uptake, by binding to and blocking the transporters. Finally, tramadol has also been shown to act as a serotonin releasing agent. Both enantiomers of tramadol are agonists of the μ-opioid receptor and its M1 metabolite, O-demethylate, which is also a μ-opioid receptor agonist but is 6 times more potent than tramadol itself. All these effects work synergistically to induce analgesia.

The aim of this study is to examine and compare the effect of both early and late intraperitoneal bupivacaine/tramadol and bupivacaine/dexmedetomedine analgesia on the effectiveness of postoperative analgesia and the requirement of postoperative rescue analgesics after laparoscopic surgery for abdominal cancer surgeries.

ELIGIBILITY:
Inclusion Criteria:

* ASA II or III.
* Age 18 to 65 years.
* Elective surgeries

Exclusion Criteria:

* Patients with severe hepatic (more than child c), renal (known CKD)and cardiac (known IHD) troubles.
* Patients with extensive intraperitoneal adhesions.
* Patients with a history of drug or analgesic abuse.
* Known drug allergy or indigestion.
* Intraoperative lavage of more than 500ml.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
The degree of pain | 24 hours
  measurement of VAS

CONTACTS AND LOCATIONS:
Overall Officials: Ehab H Gendy, MD, Principal Investigator — Assistant Professor of Anesthesia, intensive care and pain releif
Locations (1):
- National Cancer Institute, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
After manuscript approval and acceptance by a journal

REFERENCES:
- [Derived] Shaker EH, Soliman MS, Hanafy A, Elsabeeny WY. Comparative Study Between Early versus Late Intraperitoneal Administration of Either Bupivacaine/Tramadol or Bupivacaine/Dexmedetomidine for Perioperative Analgesia in Abdominal Laparoscopic Cancer Surgeries: A Prospective Randomized Study. J Pain Res. 2022 Oct 18;15:3233-3243. doi: 10.2147/JPR.S376681. eCollection 2022. PMID 36281310
- See also: Intraperitoneal dexmedetomidine as an adjuvant to bupivacaine for postoperative pain — https://www.saudija.org/article.asp?issn=1658-354X;year=2018;volume=12;issue=3;spage=399;epage=405;aulast=Elnabtity